CLINICAL TRIAL: NCT03531515
Title: Predictors of Reactive Thrombocytosis in Critically Ill Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2018-26-MD-EXP
Record Dates: First submitted 2018-03-17; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Sepsis; Thrombocytosis; Critically Ill
MeSH Terms: conditions — Sepsis; Thrombocytosis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reactive or secondary thrombocytosis is defined as abnormally high platelet count (≥4,50,000 platelets per micro-liter) in the absence of chronic myeloproliferative disease. In critically ill patients reactive thrombocytosis is not uncommon during recovery phase and an association has been seen with poor outcome and increased risk of subsequent VTE. However, not all patients with infection respond with thrombocytosis. No study has enumerated the risk factors or predictors of reactive thrombocytosis in critically ill septic patients.

DETAILED DESCRIPTION:
All patients admitted to intensive care unit of the department of Critical Care Medicine during one year period will be screened for possible inclusion in this study. In this prospective observational study, demographic and clinical characteristics of all ICU patients who fulfill inclusion criteria will be collected along with relevant laboratory tests done for patient management routinely. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Failure Assessment (SOFA) score will also be recorded. ICU survivors will be followed up in their routine ICU follow up clinic visits.

Sample size was estimated at 10% incidence rate of reactive thrombocytes, two sided 95% confidence interval and 4.5% margin of error of the incidence rate, sample size came out to be 171. Finally in this study investigators have targeted to include at least 180 participants. Sample size was estimated using software power analysis and sample size, 2008 (PASS-8).

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years) ICU patients with the diagnosis of sepsis will be considered.

Exclusion Criteria:

* Age <18 years
* Pregnancy
* H/O Malignancy
* Thrombocytosis at admission
* Primary thrombocytosis
* Post-splenectomy
* Chronic inflammatory disease (e.g. Connective tissue disorders, IBD, temporal arteritis)
* Known immunosupressive condition
* Chronic infectious diseases (e.g. tuberculosis, chronic pneumonitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) ICU patients with the diagnosis of sepsis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Reactive or secondary thrombocytosis in critically ill septic patients | From date of inclusion until the date of thrombocytosis or date of ICU discharge (death or alive), whichever came first, assessed up to 3 months
  Reactive or secondary thrombocytosis (≥4,50,000 platelets per micro-liter) due to the sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh, India